CLINICAL TRIAL: NCT01659138
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Study Evaluating Efficacy and Safety of SAR339658 in Patients With Active Moderate to Severe Ulcerative Colitis (UC)
Brief Title: Efficacy and Safety of SAR339658 in Patients With Moderate to Severe Ulcerative Colitis
Acronym: FUSCIA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment was early terminated due to slow recruitment. Not linked to any safety concern.
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACT12688; 2012-002013-19 (EudraCT Number); U1111-1124-1076 (Other: UTN)
Record Dates: First submitted 2012-08-03; First posted 2012-08-07 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SAR339658 (Experimental): SAR339658 at Weeks 0, 2, 4, and 6
  Interventions: Drug: SAR339658
- Placebo (Placebo Comparator): Placebo at Weeks 0, 2, 4, and 6
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: SAR339658 — Pharmaceutical form:solution for infusion
  Route of administration: intravenous
  Other Names: Vatelizumab
  Arms: SAR339658
Other: Placebo — Pharmaceutical form: solution for infusion
  Route of administration: intravenous
  Arms: Placebo

SUMMARY:
Primary Objective:

To assess the efficacy of SAR339658

Secondary Objective:

To assess the safety of SAR339658

DETAILED DESCRIPTION:
The study period per patient will include up to 4 weeks screening, 8 weeks treatment, 6 weeks post treatment safety follow-up, followed by a long term safety follow-up performed in the form of a phone interview at 3, 6, 12, 18 and 24 months from the last administration of the study medication.

After completion of the 8-week treatment phase, patients may be eligible to enter a long term safety study (LTS12593) for active treatment with SAR339658.

ELIGIBILITY:
Inclusion criteria:

* Male or Female ≥18 and ≤70 years old
* History of active ulcerative colitis of at least 3 months duration
* Active UC should be confirmed by colonoscopy or flexible sigmoidoscopy during the screening period within 7 days prior to randomization.
* Moderate to severe ulcerative colitis at time of screening, confirmed by Mayo score ≥6 to 12 and endoscopy subscore of ≥2 despite treatment with immunosuppressants and/or anti-tumor necrosis factors (TNFs):

  * Immunosuppressants: Patient must be on concurrent treatment with or have had an inadequate response to (did not respond to or lost response to) or be intolerant to immunosuppressants such as azathioprine, 6-mercaptopurine, or methotrexate.
  * AND/OR
  * TNF-alpha antagonists: Patient must have had an inadequate response or lost response or be intolerant to TNF-alpha antagonists
* Fecal calprotectin ≥200mg/kg
* Patients on corticosteroids must be on a stable dose ≥2 weeks prior to screening
* Patients on azathioprine, 6- mercaptopurine or methotrexate must be on treatment for at least 12 weeks prior to screening; and on a stable dose ≥4 weeks prior to screening
* Patients on oral 5-aminosalicylates, mesalamine or sulfasalazine must be on a stable dose for ≥4 weeks prior to screening
* Patients naïve to anti-TNF alpha or non-responder (primary or secondary) or intolerant to anti-TNF alpha
* Signed written informed consent

Exclusion criteria:

* Patients with Crohn's Disease
* Diagnosis of indeterminate colitis
* Patients with stool sample positive for ova, parasites, or positive culture for aerobic pathogens including: Aeromonas, Plesiomonas, Shigella, Yersinia, Campylobacter and E. Coli spp. or positive for Clostridium difficile B toxin in stools.
* Patients with prior colectomy or anticipated colectomy during their participation in the study
* Presence of ileal pouch or ostomy
* Fulminant disease or toxic megacolon
* Colonic dysplasia except for adenoma
* Total Parenteral Nutrition
* Cyclosporine, mycophenolate mofetil, sirolimus (rapamycin), thalidomide or tacrolimus within 2 months prior to screening
* Previous exposure to natalizumab (Tysabri®) or vedolizumab
* Antidiarrheals within 2 weeks prior to screening
* Prednisone >40 mg/day (or equivalent)
* Budesonide >9 mg/day
* Received intravenous corticosteroids within 2 weeks prior to screening or during screening
* Rectally administered topical 5-aminosalicylate or corticosteroids within 4 weeks prior to screening
* Received therapeutic enema or suppository, other than required for colonoscopy or flexible sigmoidoscopy within 4 weeks prior to screening or during screening
* Antibiotics for ulcerative colitis or gastrointestinal infection within 4 weeks prior to screening
* Patient who has previously participated in any clinical trial of GBR500 / SAR339658
* Patient who has taken other investigational medications within 2 months or 5 half lives, (whichever is longer) prior to screening
* Use of any biologics for the treatment of ulcerative colitis in the previous 8 weeks before screening
* Requirement for concomitant treatment that could bias primary evaluation
* Pregnant or breast-feeding women
* Women of childbearing potential not protected by highly effective contraceptive method of birth control
* Patient with latent or active tuberculosis (TB) defined as:

  * Any signs or symptoms suggestive of active TB upon medical history or clinical examination
  * Patients with a positive QuantiFERON TB Gold Test
  * Chest radiograph within 3 months prior to the inclusion visit consistent with prior tuberculosis infection including, but not limited to, apical scarring, apical fibrosis, or multiple calcified granulomasa. This does not include non-caseating granulomasa
  * Patients with close contact with a person with active tuberculosis
* Patient with a history of listeriosis or tuberculosis (unless it is documented that they were adequately treated)
* Administration of any live (attenuated) vaccine within 3 months prior to the screening Visit (eg, varicella-zoster vaccine, oral polio, rabies)
* Positive Hepatitis B surface antigen (HBsAg) or positive Hepatitis B core antibody (HBcAb); and/or positive Hepatitis C antibody (HCV) at the Screening Visit
* Prior opportunistic infections within 6 months prior to screening or while receiving anti-TNF treatment
* History of a hypersensitivity reaction, other than localized injection site reaction, to any biological molecule
* History or any current signs of demyelinating disease or any neurological disease that can by the opinion of Investigator interfere with study safety assessments including assessment for progressive multifocal leukoencephalopathy
* Patients with bleeding disorders or known platelet dysfunction

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-08; Primary Completion 2014-06 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Proportion of Participants with Clinical Response by Mayo Score | At Week 8

SECONDARY OUTCOMES:
Proportion of Participants with Clinical Remission by Mayo Score | At Week 8
Proportion of Participants with Mucosal Healing | At Week 8
Change from Baseline in Inflammatory Bowel Disease Questionnaire (IBDQ) | At Weeks 4 and 8
Change from Baseline in Quality of Life (QoL) SF-36 | At Weeks 4 and 8
Change from Baseline in the partial Mayo Score | At Weeks 4 and 6
Number of Participants with adverse events | Up to Week 17

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (41):
- United States (25):
  - Investigational Site Number 840065, Sun City, Arizona
  - Investigational Site Number 840059, Mission Hills, California
  - Investigational Site Number 840074, San Diego, California
  - Investigational Site Number 840061, Littleton, Colorado
  - Investigational Site Number 840003, Miami, Florida
  - Investigational Site Number 840008, Miramar, Florida
  - Investigational Site Number 840048, Winter Park, Florida
  - Investigational Site Number 840053, Savannah, Georgia
  - Investigational Site Number 840001, Chicago, Illinois
  - Investigational Site Number 840005, Oak Lawn, Illinois
  - Investigational Site Number 840078, Hammond, Louisiana
  - Investigational Site Number 840070, Rochester Hills, Michigan
  - Investigational Site Number 840060, Ocean Springs, Mississippi
  - Investigational Site Number 840024, Mexico, Missouri
  - Investigational Site Number 840051, Great Neck, New York
  - Investigational Site Number 840071, Rochester, New York
  - Investigational Site Number 840089, Winston-Salem, North Carolina
  - Investigational Site Number 840046, Cincinnati, Ohio
  - Investigational Site Number 840045, Phoenixville, Pennsylvania
  - Investigational Site Number 840019, Pasadena, Texas
  - Investigational Site Number 840088, San Antonio, Texas
  - Investigational Site Number 840038, Sugar Land, Texas
  - Investigational Site Number 840068, Charlottesville, Virginia
  - Investigational Site Number 840034, Seattle, Washington
  - Investigational Site Number 840064, Wauwatosa, Wisconsin
- Investigational Site Number 040003, Innsbruck, Austria
- Investigational Site Number 124002, Vancouver, Canada
- France (2):
  - Investigational Site Number 250003, Grenoble
  - Investigational Site Number 250006, Vandœuvre-lès-Nancy
- Germany (3):
  - Investigational Site Number 276001, Berlin
  - Investigational Site Number 276007, Hamburg
  - Investigational Site Number 276005, Hamburg
- Italy (2):
  - Investigational Site Number 380003, Florence
  - Investigational Site Number 380006, San Giovanni Rotondo
- Poland (7):
  - Investigational Site Number 616001, Gdynia
  - Investigational Site Number 616004, Lodz
  - Investigational Site Number 616005, Lodz
  - Investigational Site Number 616002, Lodz
  - Investigational Site Number 616007, Poznan
  - Investigational Site Number 616006, Środa Wielkopolska
  - Investigational Site Number 616008, Warsaw